CLINICAL TRIAL: NCT03114176
Title: Effects of Exercise and Dietary Inatke on Muscle Metabolism and Inflammatory Status Modulated by Oxygen Free Radicals and Cytokines in Humans
Brief Title: Effects of Ketogenic Diet in Divers Breathing Enriched Air Nitrox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Associate Professor, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NEPL-DSB 06/16
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Overweight and Obesity; Exertion; Excess; Oxygen Toxicity
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Divers group (Experimental): Throughout each dive, subjects performed a 20-minute long mild exercise on an underwater bike. The depth of dive was set at 15 meters, where the subjects performed an activity guided by Borg CR-10 scale at intensity level 3 (25 rpm). The ascent rate was set at 10 m/min, with a decompression stop at 5 meters for 3 min, according to the US Navy Manual Diving Table. 48 h prior to the immersions, none of the participants consumed medications or dived or flew. In the first part of the experiment, all subjects performed a dive breathing Enriched Air Nitrox (EAN, 32% ppO2). Baseline clinical measurements were collected before and after this first dive in order to have a reference [CTRL] and to measure physiological modifications due to immersion [NTRX]. After twenty days of no diving activity, subjects were engaged in a KD for seven days. At the end of this period, subjects performed a single immersion breathing EAN. The measures were performed after this single dive [KETO-NTRX]
  Interventions: Dietary Supplement: Ketogenic Diet

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — Diet consisted of a very low carbohydrate ketogenic diet (for 7 days) with the use of some phytoextracts as previously described. The consumed diet was primarily made of beef and veal, poultry, fish, raw and cooked green vegetables without restrictions, cold cuts (dried beef, carpaccio and cured ham), eggs and seasoned cheese (e.g., parmesan). The allowed drinks were infused tea, moka coffee and herbal extracts. The foods and drinks that subjects had to avoid included alcohol, bread, pasta, rice, milk, yogurt, soluble tea, and barley coffee. To facilitate adherence to the nutritional regime, a variety of special meals based on protein and fibers were given to each subject. KD characteristics are protein intake 1.3g/kg/day, to maintain skeletal muscle mass; carbohydrates intake less than 40 g/day and 50-60% of total kcal to induce ketosis. In accordance with a hypocaloric profile, total energy intake was calculated with 200 kcal more than basal metabolic rate.

SUMMARY:
Overweight divers face a challenging activity such as immersions, starting from a higher levels of circulating cytokines and oxidative stress. Ketogenic Diet (KD) is described as effective in weight loss, in countering inflammation and oxidative stress, and used in the control of drug-refractory seizures.

The aim of our pilot study was to evaluate if a ketosis state induced by a specific dietary regime, may have a protective effect on oxidative stress damages and inflammatory status, that accompanies both overweight and diving activities.

Blood and urine samples from six overweight divers were obtained a) before (CTRL) and after a dive breathing Enriched Air Nitrox and performing light underwater exercise (NTRX), b) after a dive (same conditions) performed after 7 days of KD (K-NTRX). We measured urinary 8-isoprostane and 8-OH-2-deoxyguanosine evaluating lipids peroxidation and DNA oxidative damages. Plasmatic IL-1beta, IL-6 and TNF-alpha levels were measured to investigate the inflammatory status.

ELIGIBILITY:
Inclusion Criteria:

* to be in an overweight state (BMI ≥ 25 kg/m2) and no history of orthopedic, cardiovascular, renal or metabolic disorders.

Exclusion Criteria:

* not to be in an overweight state (BMI ≥ 25 kg/m2) and a history of orthopedic, cardiovascular, renal or metabolic disorders.

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05-25 (Actual); Primary Completion 2016-07-10 (Actual); Study Completion 2016-07-10 (Actual)

PRIMARY OUTCOMES:
Oxidative damage change | Change from Baseline Oxidative damage at twenty days
  8-OH-dG (ng ⋅ mg-1 creatinine) and 8-iso-PGF2α (ng ⋅ mg-1 creatinine)
Pro-inflammatory cytokines change | Change from Baseline Pro-inflammatory cytokines at twenty days
  IL-1β (pg/ml), IL-6 (pg/ml) and TNF- α (pg/ml)

SECONDARY OUTCOMES:
Weight Loss | Weight was registered before (T0) and after twenty days of no diving activity in which subjects were engaged in a 7-days Ketogenic Diet (T3).
  Kilogram (Kg)

CONTACTS AND LOCATIONS:
Overall Officials: Bosco Gerardo, MD, PhD, Study Director — University of Padova

IPD SHARING:
Plan to Share IPD: No